CLINICAL TRIAL: NCT02260791
Title: A Randomised, Blinded, Active-Controlled Study to Compare FKB327 Efficacy and Safety With the Comparator Humira® in Rheumatoid Arthritis Patients Inadequately Controlled on Methotrexate
Brief Title: A Study to Compare FKB327 Efficacy and Safety With Humira® in Rheumatoid Arthritis Patients
Acronym: ARABESC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujifilm Kyowa Kirin Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FKB327-002
Record Dates: First submitted 2014-07-29; First posted 2014-10-09 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — FKB327; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FKB327 (Experimental): Patients will receive FKB327 40 mg every other week by subcutaneous injection. The treatment period will continue for 22 weeks.
  Interventions: Drug: FKB327
- Humira® (Active Comparator): Patients will receive Humira® 40 mg every other week by subcutaneous injection. The treatment period will continue for 22 weeks.
  Interventions: Drug: Humira®

INTERVENTIONS:
Drug: FKB327 — Solution of FKB327 for subcutaneous injection administered in a dose of 40 mg every 2 weeks for 22 weeks.
  Arms: FKB327
Drug: Humira® — Solution of Humira® for subcutaneous injection administered in a dose of 40 mg every 2 weeks for 22 weeks.
  Arms: Humira®

SUMMARY:
The purpose of the study is to compare the effectiveness and safety of FKB327 in comparison to Humira® in rheumatoid arthritis patients who have inadequate disease control on methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or over
2. Patients have been diagnosed with Rheumatoid Arthritis (RA) for at least 3 months
3. Patient has active RA
4. Patient has taken a stable dose of methotrexate for at least 3 months

Exclusion Criteria:

1. Patient has been previously treated with adalimumab
2. Patient has been previously treated or has ongoing treatment with prohibited medications
3. Patient has been immunised with a live or attenuated vaccine in past 4 weeks
4. Patient has positive result for HIV, HBV, HCV or TB infection

Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Glover, MD, Principal Investigator — Coephycient Pharmaceutical Consultancy
Locations (100):
- United States (16):
  - Research Site, Peoria, Arizona
  - Research Site, Palm Desert, California
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Lansing, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Mesquite, Texas
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (3):
  - Research Site, Mississauga, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Trois-Rivières, Quebec
- Chile (5):
  - Research Site, Osorno
  - Research Site, Puerto Varas
  - Research Site G, Santiago
  - Research Site M, Santiago
  - Research Site, Temuco
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hlučín
  - Research Site U, Prague
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Germany (6):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Hildesheim
  - Research Site, Munich
  - Research Site, Ratingen
- Peru (7):
  - Research Site B, Arequipa
  - Research Site M, Arequipa
  - Research Site CA, Lima
  - Research Site CH, Lima
  - Research Site PA, Lima
  - Research Site PE, Lima
  - Research Site S, Lima
- Poland (10):
  - Research Site D, Bialystok
  - Research Site R, Bialystok
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site KL, Krakow
  - Research Site KR, Krakow
  - Research Site, Lublin
  - Research Site P, Poznan
  - Research Site RH, Poznan
  - Research Site, Torun
- Romania (9):
  - Research Site, Oradea, Bihor County
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site C, Bucharest
  - Research Site R, Bucharest
  - Research Site T, Bucharest
  - Research Site, Constanța
  - Research Site, Galati
  - Research Site, Sfântu Gheorghe
- Russia (17):
  - Research Site, Ufa, Bashkortostan Republic
  - Research Site, Petrozavodsk, Karelia Republic
  - Research Site, Kazan', Tatarstan Republic
  - Research Site D, Moscow
  - Research Site SM, Moscow
  - Research Site ST, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site B, Saint Petersburg
  - Research Site Z, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Vladimir
  - Research Site E, Yaroslavl
  - Research Site S, Yaroslavl
- Spain (5):
  - Research Site, Santiago de Compostela, La Coruna
  - Research Site, Bilbao, Vizcaya
  - Research Site A, Barcelona
  - Research Site G, Barcelona
  - Research Site, Málaga
- Ukraine (14):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site A, Kyiv
  - Research Site B, Kyiv
  - Research Site P, Kyiv
  - Research Site, Lutsk
  - Research Site C, Lviv
  - Research Site N, Lviv
  - Research Site, Poltava
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site G, Vinnytsia
  - Research Site Sh, Vinnytsia
  - Research Site St, Vinnytsia

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Genovese MC, Glover J, Greenwald M, Porawska W, El Khouri EC, Dokoupilova E, Vargas JI, Stanislavchuk M, Kellner H, Baranova E, Matsunaga N, Alten R. FKB327, an adalimumab biosimilar, versus the reference product: results of a randomized, Phase III, double-blind study, and its open-label extension. Arthritis Res Ther. 2019 Dec 12;21(1):281. doi: 10.1186/s13075-019-2046-0. PMID 31831079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 109 sites in 12 countries in 3 geographical regions: North America, Europe and Rest of World. The first participant enrolled on 05 January 2015 and the last participant completed on 12 July 2016.
Pre-assignment Details: Screening details:
  Patients were randomised in a 1:1 ratio to receive either FKB327 40 mg eow or Humira 40 mg eow using the following stratification factors: prior biological treatment for Rheumatoid Arthritis (RA) (yes/no) and Screening disease activity (DAS28-CRP ≤5.1/>5.1).
Groups:
- FKB327: Patients were administered subcutaneous (sc) FKB327 40 mg every other week (eow). The treatment period was 22 weeks.
- Humira®: Patients were administered subcutaneous (sc) Humira 40 mg every other week (eow). The treatment period was 22 weeks.
Period: Overall Study
Arm/Group | FKB327 | Humira®
Started | 366 | 362
Completed | 333 | 328
Not Completed | 33 | 34
Not completed — Lost to Follow-up | 4 | 4
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 13 | 9
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 11 | 16
Not completed — Screen failure | 0 | 1
Not completed — Protocol deviation | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was defined as the set of patients who received at least 1 dose of randomised treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | FKB327 | Humira® | Total
Number analyzed (Participants) | 366 | 362 | 728
Age, Continuous [Mean (Full Range); unit: years] | 53 [18 to 85] | 53.6 [21 to 93] | 53.3 [18 to 93]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 65 years | 302 | 299 | 601
  >65 years | 64 | 63 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 284 | 565
  Male | 85 | 78 | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 311 | 308 | 619
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 51 | 48 | 99
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 4 | 7
  Romania | 15 | 13 | 28
  United States | 39 | 39 | 78
  Czech Republic | 33 | 34 | 67
  Ukraine | 56 | 58 | 114
  Poland | 67 | 67 | 134
  Bulgaria | 7 | 7 | 14
  Chile | 20 | 21 | 41
  Peru | 51 | 49 | 100
  Germany | 14 | 12 | 26
  Spain | 4 | 6 | 10
  Russia | 57 | 52 | 109

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response Rate
Description: The primary efficacy endpoint was the ACR20 response rate at Week 24.
  An ACR20 response meant that the patient achieved a 20% improvement in Tender Joint Count and Swollen Joint Count and in at least 3 of the other 5 Core Data Set elements listed below.
  * Acute phase reactant (CRP)
  * Patient global assessment of disease activity
  * Physician global assessment of disease activity
  * Patient pain scale
  * Disability/functional questionnaire (patient completed Health Assessment Questionnaire Disability Index [HAQ-DI])
Time Frame: Week 24
Population: The Full Analysis Set (FAS) was defined as the set of patients who received at least 1 dose of the randomised treatment and who had at least 1 evaluable primary efficacy measurement after their first dose of randomised treatment. Patients were analysed according to the randomised treatment in the primary analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
Percentage of participants | 72.5 [67.5 to 77.0] | 74.3 [69.4 to 78.8]
Statistical Analysis 1: Comparison: FKB327 vs Humira®; The difference and its 90% Confidence Interval (CI) for primary endpoint between FKB327 and Humira were estimated. If the 90% CI fell entirely between pre-specified equivalence margin (-12% to +15%), then FKB327 was considered equivalent to Humira; Test type: Equivalence — -12% to +15% equivalence margin using 90% CI around the difference in ACR20 response rate; Mean Difference (Final Values) = -1.8, 90% CI 2-sided [-7.3 to 3.6]

2. Secondary Outcome: Disease Activity Score 28 (DAS28) Based on C-reactive Protein (DAS28-CRP) Score
Description: The DAS28-CRP assessment involved evaluating the number of tender (TJC) and swollen (SJC) joints (out of 28 specified joints), serum CRP, and patient global assessment of disease activity (VAS from 0 to 100, very well to extremely bad). The DAS28-CRP is a number on a scale from 0 to 10 indicating the current activity of the patient's RA. A higher score indicates higher disease activity.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline: number analyzed (Participants) | 362 | 358
  Baseline | 6.05 (0.913) | 6.06 (0.852)
  Week 2: number analyzed (Participants) | 361 | 351
  Week 2 | 4.92 (1.070) | 4.86 (1.203)
  Week 4: number analyzed (Participants) | 357 | 348
  Week 4 | 4.44 (1.317) | 4.43 (1.383)
  Week 8: number analyzed (Participants) | 348 | 345
  Week 8 | 4.11 (1.295) | 4.09 (1.397)
  Week 12: number analyzed (Participants) | 351 | 340
  Week 12 | 3.81 (1.320) | 3.85 (1.339)
  Week 16: number analyzed (Participants) | 350 | 341
  Week 16 | 3.68 (1.304) | 3.67 (1.419)
  Week 20: number analyzed (Participants) | 344 | 336
  Week 20 | 3.58 (1.329) | 3.57 (1.388)
  Week 24: number analyzed (Participants) | 340 | 339
  Week 24 | 3.47 (1.298) | 3.47 (1.336)
Statistical Analysis 1: Comparison: FKB327 vs Humira®; The secondary hypothesis involved equivalence of the difference between FKB327 and Humira in DAS28-CRP at Week 24. Based on the repeated measures analysis model, the difference and its 95% CI in the least-squares means (LSMs) for DAS28-CRP at Week 24 between FKB327 and Humira were estimated. If the 95% CI fell entirely between the pre-specified margin (+/- 0.6), then FKB327 was considered equivalent to Humira; Test type: Equivalence — If the 2-sided 95% CI for the difference in DAS28-CRP at Week 24 between FKB327 and Humira fell entirely between -0.6 and +0.6 then FKB327 was considered equivalent to Humira; Difference in least square mean = 0.01, 95% CI 2-sided [-0.16 to 0.18]

3. Secondary Outcome: ACR20 Response Rates Over Time
Description: An ACR20 response meant that the patient achieved a 20% improvement in Tender Joint Count and Swollen Joint Count and in at least 3 of the other 5 Core Data Set elements listed below.
  * Acute phase reactant (CRP)
  * Patient global assessment of disease activity
  * Physician global assessment of disease activity
  * Patient pain scale
  * Disability/functional questionnaire (patient completed Health Assessment Questionnaire Disability Index [HAQ-DI])
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: The Full Analysis Set (FAS) was defined as the set of patients who received at least 1 dose of the randomised treatment and who had at least 1 evaluable primary efficacy measurement after their first dose of randomised treatment.Patients were analysed according to the randomised treatment in the primary analysis.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
percentage of responders
  Week 2: number analyzed (Participants) | 362 | 352
  Week 2 | 37.3 [32.3 to 42.5] | 31 [26.2 to 36.1]
  Week 4: number analyzed (Participants) | 359 | 349
  Week 4 | 51 [45.7 to 56.3] | 52.4 [47.1 to 57.8]
  Week 8: number analyzed (Participants) | 353 | 347
  Week 8 | 64.6 [59.4 to 69.6] | 67.7 [62.5 to 72.6]
  Week 12: number analyzed (Participants) | 351 | 342
  Week 12 | 69.2 [64.1 to 74] | 72.2 [67.2 to 76.9]
  Week 16: number analyzed (Participants) | 350 | 342
  Week 16 | 74.6 [69.7 to 79.1] | 74.9 [69.9 to 79.4]
  Week 20: number analyzed (Participants) | 345 | 338
  Week 20 | 78 [73.2 to 82.2] | 77.8 [73 to 82.1]
  Week 24: number analyzed (Participants) | 341 | 338
  Week 24 | 77.1 [72.3 to 81.5] | 79.3 [74.6 to 83.5]

4. Secondary Outcome: ACR50 Response Rates Over Time
Description: An ACR50 response meant that the patient achieved a 50% improvement in Tender Joint Count and Swollen Joint Count and in at least 3 of the other 5 Core Data Set elements listed below.
  * Acute phase reactant (CRP)
  * Patient global assessment of disease activity
  * Physician global assessment of disease activity
  * Patient pain scale
  * Disability/functional questionnaire (patient completed Health AssessmentQuestionnaire Disability Index [HAQ-DI])
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
percentage of responders
  Week 2: number analyzed (Participants) | 362 | 352
  Week 2 | 5 [3 to 7.7] | 8.8 [6.1 to 12.3]
  Week 4: number analyzed (Participants) | 359 | 349
  Week 4 | 17.3 [13.5 to 21.6] | 17.8 [13.9 to 22.2]
  Week 8: number analyzed (Participants) | 353 | 346
  Week 8 | 28.9 [24.2 to 33.9] | 30.9 [26.1 to 36.1]
  Week 12: number analyzed (Participants) | 351 | 342
  Week 12 | 37.6 [32.5 to 42.9] | 35.1 [30 to 40.4]
  Week 16: number analyzed (Participants) | 350 | 342
  Week 16 | 39.4 [34.3 to 44.8] | 44.7 [39.4 to 50.2]
  Week 20: number analyzed (Participants) | 345 | 339
  Week 20 | 45.5 [40.2 to 50.9] | 46 [40.6 to 51.5]
  Week 24: number analyzed (Participants) | 341 | 338
  Week 24 | 49 [43.6 to 54.4] | 49.4 [44 to 54.9]

5. Secondary Outcome: ACR70 Response Rates Over Time
Description: An ACR70 response meant that the patient achieved a 70% improvement in Tender Joint Count and Swollen Joint Count and in at least 3 of the other 5 Core Data Set elements listed below.
  * Acute phase reactant (CRP)
  * Patient global assessment of disease activity
  * Physician global assessment of disease activity
  * Patient pain scale
  * Disability/functional questionnaire (patient completed Health AssessmentQuestionnaire Disability Index [HAQ-DI])
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
percentage of responders
  Week 2: number analyzed (Participants) | 362 | 352
  Week 2 | 0.3 [0 to 1.5] | 2.3 [1 to 4.4]
  Week 4: number analyzed (Participants) | 359 | 349
  Week 4 | 4.5 [2.6 to 7.1] | 6.9 [4.5 to 10.1]
  Week 8: number analyzed (Participants) | 353 | 347
  Week 8 | 11.3 [8.2 to 15.1] | 10.7 [7.6 to 14.4]
  Week 12: number analyzed (Participants) | 351 | 342
  Week 12 | 15.4 [11.8 to 19.6] | 13.2 [9.8 to 17.2]
  Week 16: number analyzed (Participants) | 350 | 342
  Week 16 | 17.4 [13.6 to 21.8] | 19 [15 to 23.6]
  Week 20: number analyzed (Participants) | 345 | 339
  Week 20 | 20.9 [16.7 to 25.5] | 23.6 [19.2 to 28.5]
  Week 24: number analyzed (Participants) | 342 | 338
  Week 24 | 21.3 [17.1 to 26.1] | 25.1 [20.6 to 30.1]

6. Secondary Outcome: Swollen Joint Count
Description: Counts of swollen joints from amongst 66 selected joints performed by a trained and qualified joint assessor using standardised techniques recommended by the European League Against Rheumatism (EULAR). Joints were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66 with higher scores indicating severe disease. Swollen joint count is a value of the individual ACR core set variables.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count / Score
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
Count / Score
  Baseline | 16.3 (9.1) | 16 (8.96)
  Week 24 | 3.8 (6.04) | 3.5 (5.23)

7. Secondary Outcome: Tender Joint Count
Description: Counts of tender joints from amongst 68 selected joints were performed by a trained and qualified joint assessor using standardised techniques recommended by the European League Against Rheumatism (EULAR). Joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68 with higher scores indicating severe disease.Tender joint count is a value of the individual ACR core set variables.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count / Score
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
Count / Score
  Baseline | 26.2 (14.49) | 25.9 (14.52)
  Week 24 | 8.5 (10.56) | 8.1 (9.36)

8. Secondary Outcome: Analysis of Serum C-Reactive Protein (CRP) Concentration
Description: Analysis of serum C-Reactive Protein (CRP) concentrations for inclusion in the ACR20/50/70 and DAS28-CRP scores was performed by a central laboratory. Elevation of CRP is a nonspecific marker of inflammation. Values above 10 mg/L were considered to be abnormally high. Decrease in level of CRP indicates reduction in inflammation.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
mg/L
  Baseline | 25.12 (26.746) | 26.73 (28.534)
  Week 24 | 10.98 (16.819) | 11.78 (18.528)

9. Secondary Outcome: Patient Assessment of Disease Activity
Description: Patient assessment of disease activity visual analogue scale (VAS) will be assessed on 100-point scales (ranging from very well (0) to extremely bad (100)).The patient assessment of disease activity VAS will contribute to the calculation of the DAS28 score. The patient assessment of disease activity VAS will contribute to the calculation of ACR20, ACR50 and ACR70 response.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline | 68 (17.98) | 68.2 (18.18)
  Week 24 | 35.2 (24.04) | 33.2 (23.4)

10. Secondary Outcome: Physician Assessment of Disease Activity
Description: Physician assessment of disease activity visual analogue scale (VAS) will be assessed on 100-point scale (ranging from very low (0) to very high (100)). The physician assessment of disease activity VAS will contribute to the calculation of ACR20, ACR50 and ACR70 response.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline | 68.4 (14.58) | 66.2 (15.48)
  Week 24 | 21.5 (17.29) | 21.5 (16.97)

11. Secondary Outcome: Patient's Assessment of Pain
Description: An injection site pain visual analogue score (VAS) will be administered to the patient. To determine the extent of the pain, patients will be asked to place a small vertical mark on a horizontal scale from 0 to 100, the ends of which are labelled with the extreme responses to be measured ("No pain" at 0 and "Intolerable pain" at 100). Patient's assessment of pain is a value of the individual ACR core set variables.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline | 66.8 (18.71) | 67.7 (18.56)
  Week 24 | 34.7 (23.86) | 33.6 (23.86)

12. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI is a 20-question, self-administered instrument that measures the patient's functional ability on a 4-level difficulty scale (0 to 3, with 0 representing normal or no difficulty and 3 representing inability to perform). Eight categories of functioning are included: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. This scale is sensitive to change and is a good predictor of future disability. HAQ-DI is a value of the individual ACR core set variables.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline | 1.78 (0.544) | 1.8 (0.538)
  Week 24 | 1.21 (0.696) | 1.26 (0.719)

13. Secondary Outcome: DAS28-CRP Score Over Time
Description: The DAS28 score is a combined index that has been developed to measure the disease activity in patients with RA and has been extensively validated for its use in clinical studies. The DAS28-CRP assessment involved evaluating the number of tender (TJC) and swollen (SJC) joints (out of 28 specified joints), serum CRP, and patient global assessment of disease activity (VAS from 0 to 100, very well to extremely bad). The individual results are summed using a formula. The DAS28 is a number on a scale from 0 to 10 indicating the current activity of the patient's RA. A higher score indicates higher disease activity.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline: number analyzed (Participants) | 362 | 358
  Baseline | 6.05 (0.913) | 6.06 (0.852)
  Week 24: number analyzed (Participants) | 340 | 339
  Week 24 | 3.47 (1.298) | 3.47 (1.336)

14. Secondary Outcome: DAS28 Score Based on Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The DAS28 score is a combined index that has been developed to measure the disease activity in patients with RA and has been extensively validated for its use in clinical studies. The DAS28-ESR assessment involved evaluating the number of tender (TJC) and swollen (SJC) joints (out of 28 specified joints), serum ESR, and patient global assessment of disease activity (VAS from 0 to 100, very well to extremely bad). The individual results are summed using a formula. The DAS28 is a number on a scale from 0 to 10 indicating the current activity of the patient's RA. A higher score indicates higher disease activity.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 363 | 358
units on a scale
  Baseline: number analyzed (Participants) | 361 | 355
  Baseline | 6.52 (0.941) | 6.56 (0.902)
  Week 12: number analyzed (Participants) | 349 | 340
  Week 12 | 4.24 (1.382) | 4.24 (1.353)
  Week 24: number analyzed (Participants) | 342 | 338
  Week 24 | 3.82 (1.384) | 3.85 (1.371)

15. Other Pre Specified Outcome: Percentage of Patients Developing Anti-drug Antibodies (ADAs)
Description: Blood samples for the assessment of ADA activity were collected at Baseline (Week 0), prior to dosing at Weeks 2, 4, 12, and 24.
Time Frame: Baseline and last sampling day
Population: The Safety Analysis Set was defined as the set of patients who received at least 1 dose of randomised treatment. The Safety Analysis Set was used for all safety analyses. Patient safety data were analysed according to treatment actually received.
Measure: Number; unit: percentage of patients
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 366 | 362
percentage of patients
  Baseline (Positive) | 4.4 | 5.5
  Baseline (Negative) | 95.4 | 94.2
  Baseline (Missing) | 0.3 | 0.3
  Last sampling day (Positive) | 61.7 | 59.1
  Last sampling day (Negative) | 38.3 | 40.9

16. Other Pre Specified Outcome: Trough Adalimumab Concentration
Description: Blood samples for the quantification of adalimumab concentration in serum were collected at Baseline (Week 0), prior to dosing at Weeks 2, 4, 12 and 20, and Week 24. Samples were taken prior to dosing (trough samples).
Time Frame: Week 2, Week 4, Week 12, Week 20, and Week 24
Population: The Pharmacokinetic Analysis Set (PKAS) was defined as the set of patients who received at least 1 dose of the randomised treatment and had at least 1 serum adalimumab concentration result after receiving randomised treatment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | FKB327 | Humira®
Number analyzed (Participants) | 364 | 358
ng/mL
  Week 2 | 2434.6 [2321.4 to 2553.2] | 2089.1 [1990.9 to 2192.2]
  Week 4 | 3450.6 [3223.2 to 3694.1] | 2932.1 [2737 to 3141.1]
  Week 12 | 4316.3 [3919.6 to 4753.2] | 3851.5 [3493.9 to 4245.7]
  Week 20 | 4369.8 [3892.3 to 4905.9] | 3873 [3445.9 to 4353]
  Week 24 | 4126 [3645.1 to 4670.4] | 3758.2 [3316.8 to 4258.3]

ADVERSE EVENTS:
Time Frame: Patients were carefully monitored for adverse events from signing of informed consent until Week 24 (for patients who entered the open-label extension), Week 26 (for patients who did not enter the open-label extension), or the Early Termination visit. In total this covered a period of approximately 1 year and 6 months.
Description: Serious adverse events were followed until resolution, the Investigator confirmed the event was unlikely to resolve or the patient was recorded as lost to follow-up.
Arm/Group | FKB327 | Humira®
All-Cause Mortality (participants affected / at risk) | 1/366 | 0/362
Serious Adverse Events (participants affected / at risk) | 15/366 | 19/362
Other Adverse Events (participants affected / at risk) | 26/366 | 29/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB327 (N=366) | Humira® (N=362)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB327 (N=366) | Humira® (N=362)
Nasopharyngitis (Infections and infestations) | 26 (26) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Sponsor will discuss the preparation of a manuscript for publication in a peer reviewed journal or an abstract for presentation. Either party may undertake the task but both must agree to the strategy before work is started. Each party will allow the other 30 days to comment before any results are submitted for publication or presentation. Authorship should reflect work done by the Investigators and Sponsor, in accordance with recognised principles of scientific collaboration.